CLINICAL TRIAL: NCT05598437
Title: Search Protocol 1. Study a-Proposed Study Title: Prevalence of Different Etiologies of Ocular Dryness in Patients Previously Diagnosed With Dry Eye Disease in A Sample of Egyptian Patients
Brief Title: Prevalence of Different Etiologies of Ocular Dryness in Patients Previously Diagnosed With Dry Eye Disease in A Sample of Egyptian Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Roweis adel youssef (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Roweis adel youssef, Cairo university, Cairo University
Organization: Cairo University (Other)
Other Study IDs: 1298756727278
Record Dates: First submitted 2022-10-25; First posted 2022-10-28 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Dryness; Dry Eye Syndromes; Meibomian Gland Dysfunction
Keywords: Dry eye disease
MeSH Terms: conditions — Dry Eye Syndromes; Meibomian Gland Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- A: Left eye
  Interventions: Device: Dry eye device
- B: Right eye
  Interventions: Device: Dry eye device

INTERVENTIONS:
Device: Dry eye device — Dry eye analysis

SUMMARY:
Proposed Study Title: Prevalence of Different Etiologies of Ocular Dryness in Patients Previously Diagnosed with Dry Eye

DETAILED DESCRIPTION:
Dry eye disease (DED) is a common chronic multifactorial condition of the ocular surface characterized by failure to produce high quality or sufficient amounts of tears to moisturize the eyes (1) DED can be categorized as "dry eye with reduced tear production (aqueous deficient) and dry eye with increased evaporation of the tear film known as the hyperevaporative type… Although 10% of individuals have aqueous deficient DED, more than 80% have either the hyperevaporative type related to meibomian gland dysfunction (MGD), or a combination of

ELIGIBILITY:
Inclusion Criteria:

* Egyptian people between 20 and 70 years old coming to outpatient clinic BUT< 10 seconds.. No previous surgery. No previous trauma. Not using eye drops in the last 3 months.

Exclusion Criteria:

Diabetic patients. Patients with rheumatological diseases that may affect ocular surface as RA.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Egyptian people between 20 and 70 years old coming to outpatient clinic BUT< 10 seconds.. No previous surgery. No previous trauma. Not using eye drops in the last 3 months.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Meibomian gland dysfunction | 6 months
  Meibomian gland dysfunction

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Study will be in6 months